CLINICAL TRIAL: NCT05396209
Title: Multicenter Case Control Clinical Trials to Compare the Healing Process of Refractory Macular Hole With Different Surgical Techniques
Brief Title: To Evaluate the Therapeutic Efficacy of Hydrated Amniotic Membrane in Promoting Closure of Refractory Macular Holes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oriental Neurosurgery Evidence-Based-Study Team (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMMH2022
Record Dates: First submitted 2022-05-24; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Macular Holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydrated Amniotic Membrane Plug (Active Comparator): Patients suffering from refractory macular holes as documented by spectral-domain OCT will undergo pars plan vitrectomy with Hydrated Amniotic Membrane insertion into the macular hole.
  Interventions: Procedure: Hydrated Amniotic Membrane Plug
- ILM filling (Active Comparator): The ILM filling technique, in which free ILM is plug into the macular hole area
  Interventions: Procedure: ILM filling
- Conventional ILM peeling (Active Comparator): Peeling with complete removal of the internal limiting membrane within the vascular arch
  Interventions: Procedure: Conventional ILM peeling

INTERVENTIONS:
Procedure: Hydrated Amniotic Membrane Plug — Using Hydrated Amniotic Membrane plug with vitrectomy to try to close refractory macular hole
  Arms: Hydrated Amniotic Membrane Plug
Procedure: ILM filling — The ILM filling technique - Rossi et al show that ILM filling technique was more efficacious in closing full-thickness macular holes larger than 630μm, in which the free ILM after peeling is plug into the area of the macular hole
  Arms: ILM filling
Procedure: Conventional ILM peeling — Peeling with complete removal of the internal limiting membrane within the vascular arch
  Arms: Conventional ILM peeling

SUMMARY:
To compare anatomic and functional results, and to evaluate postoperatively the healing process in 3 different techniques for the closure of the refractory macular holes (MH).

DETAILED DESCRIPTION:
The aim of the study is to evaluate the therapeutic efficacy of Hydrated Amniotic Membrane in promoting closure of refractory macular holes.

The Hydrated Amniotic Membrane has been used in some cases as an adjunct in the macular holes closure and as a substrate for cell growth and improvement of visual acuity. Hydrated Amniotic Membrane is supposed to promote epithelialization and have anti-fibrotic, anti-inflammatory properties.

In the present study, the patients who meet the inclusion criteria will be randomized and undergo pars plana vitrectomy surgery with peeling of the ILM and a fragment of the ILM itself or an amniotic membrane plug will be put in place.

The patients included in the study will undergo a complete eye examination, including corrected Visual Acuity measurement (BCVA), performing the Optical Coherence Tomography (OCT) and/or microperimetry, multifocal electroretinogram (mfERG) in the pre-operative. Patients will undergo surgery after complementary exams and adequate pre-anesthetic evaluation.

Patients will be evaluated on the 1st and 7th postoperative days and at 1, 3, and 6 months after surgery. The patient will undergo a complete eye examination and postoperative follow-up as described above, and during visits on the 1st and 7th day, and in the 1st, 3th and 6th month of the postoperative period, BCVA and OCT will be performed and/or the microperimetry, multifocal electroretinogram (mfERG) will be performed in the 1st, 3th and 6th postoperative month for evaluation and monitoring of anatomical and functional responses, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. idiopathic macular hole was defined as macular hole diameter (with no history of secondary macular hole) larger than 800μm in minimum linear diameter ;
2. Patients with an idiopathic macular hole submitted to pars plana vitrectomy with internal limiting membrane peeling treatment without closing it and macular hole diameter larger than 200μm.

Patients who meet any of 1/2 and signed informed consent can be included. Note: if both eyes of the subject meet the inclusion criteria, the investigator decides which eye should be included.

Exclusion Criteria:

1. idiopathic macular hole diameter less than 800μm in minimum linear diameter;
2. Macular hole caused by trauma and laser;
3. Macular holes secondary to another vitreoretinal diseases;
4. Macular hole of pathological myopia (axial length ≥26.0mm and diopter ≥6.00D，posterior scleral staphyloma，the atrophic choroid and retina with scleral exposure);
5. Known to be allergic to amniotic membrane.

   Patients with any of the following eye diseases:
6. Patients with other ocular disease (diabetic retinopathy, glaucoma, uveitis, ocular tumors, etc);
7. Macular hole of other causes (secondary)；
8. History of vitreoretinal surgery for a condition other than the idiopathic macular hole (retinal detachment, vitreous hemorrhage);

   Patients with any of the following eye conditions:
9. Using systemic drugs that are toxic for the optic nerve or retina (chloroquine, hydroxychloroquine, tamoxifen, ethambutol, etc)；
10. Patients with ocular surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Rate of Anatomic closure | Month 6 post operative
  Rate of anatomic macular hole closure in the OCT at month 6
Reconstruction of the foveal layered retinal structure change | Month 1, 3, 6 post-operative
  Change in the reconstruction of the foveal layered retinal structure by OCT at 1, 3, and 6 months

SECONDARY OUTCOMES:
amniotic membrane dislocation | DAY 1,7 post operative
  conform amniotic membrane dislocation in the OCT and/or binocular indirect ophthalmoscope at day 1 and 7
BCVA change | Time Frame: Preoperative,Month 1, 3, 6 post operative
  change in the BCVA at Preoperative,1, 3, and 6 months
Retinal capillary plexus density change | Preoperative,Month 1, 3, 6 post operative
  change in the retinal capillary plexus density with OCT-A at Preoperative,1, 3, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hua Yan, MD,PhD, Principal Investigator — Ophthalmology of Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China